CLINICAL TRIAL: NCT03479502
Title: Intra-articular Doxycycline: A Novel Treatment of Adhesive Capsulitis
Acronym: DOXY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Principal Investigator, John Kuhn, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 172011
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Adhesive Capsulitis; Adhesive Capsulitis of Unspecified Shoulder; Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Prednisone; Doxycycline

STUDY DESIGN:
Intervention Model Description: Patients meeting the inclusion criteria will be randomized into either the control group of intra-articular injection of 40mg Methylprednisolone once every 2 two weeks for 4 weeks (day 1, week 2, week 4) or the experimental group of intraarticular injection of 50 mg doxycycline once every 2 two weeks for 4 weeks (day 1, week 2, week 4), with 20 patients in each group. Injections will be administered by the treating physician. The Vanderbilt Investigational Pharmacy will provide the doxycycline and the steroid solutions and will be in charge of patient randomization.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone (Active Comparator): Patients meeting the inclusion criteria will be randomized into either the control group of intra-articular injection of 40mg Methylprednisolone once every 2 two weeks for 4 weeks (day 1, week 2, week 4) with 20 patients in each group. Injections will be administered by the treating physician.
  Interventions: Drug: Methylprednisolone Injectable Product
- Doxycycline (Active Comparator): Patients meeting the inclusion criteria will be randomized or the experimental group of intraarticular injection of 50 mg doxycycline once every 2 two weeks for 4 weeks (day 1, week 2, week 4), with 20 patients in each group. Injections will be administered by the treating physician.
  Interventions: Drug: Doxycycline Injection

INTERVENTIONS:
Drug: Methylprednisolone Injectable Product — 3 intra-articular injections of Methylprednisolone Injectable Product spaced every two weeks
  Other Names: Prednisone
  Arms: Methylprednisolone
Drug: Doxycycline Injection — 3 intra-articular injections of Doxycycline Injection spaced every two weeks
  Other Names: Doxy
  Arms: Doxycycline

SUMMARY:
We will recruit a total of 40 patients from the Vanderbilt Sports Medicine Clinics who have been diagnosed with adhesive capsulitis and have not undergone any previous treatment. The 40 patients will be randomized, with 20 in the control group of 3 intra-articular injections of 40mg Methylprednisolone spaced every two weeks, and 20 in the experimental group of 3 intra-articular injection of 50mg doxycycline spaced every two weeks. Both groups will begin a standardized physical therapy program within a pain-free range of motion 4 weeks after the initiation of treatment. We will prospectively follow patients for one year, with follow-up at 6 weeks, 12 weeks, 6 months, and 12 months after the initiation of treatment.

Outcomes will be measured using the American Shoulder and Elbow Score (ASES) and objective measurements of shoulder range of motion, which will be collected by the treating physician. Both the patients and physicians participating in the study will be blinded.

DETAILED DESCRIPTION:
Adhesive capsulitis, also known as frozen shoulder, is a common condition of the shoulder joint affecting 2-5% of the adult population and characterized by progressive, painful loss of both passive and active range of motion of shoulder [1,2]. Individuals affected by this condition find it increasingly difficult to perform activities of daily living that require overhead movement or rotation of the affected shoulder. The natural history of frozen shoulder follows a predictable progression of symptoms, lasting from 9-24 months before complete resolution, and results in significant loss of productivity and quality of life for those affected [3]. Despite the significant number of patients affected by adhesive capsulitis and the extensive literature focused on the progression and natural history of the condition, the true underlying etiology remains poorly understood. In light of this poor understanding of the condition, it is not surprising that a number of conservative and invasive modalities exist as accepted treatments. These include non-steroidal anti-inflammatory drugs (NSAIDS), oral steroids, intra-articular steroid injections, Physical Therapy (PT), and benign neglect as well as more invasive treatments such as hydroxylation, manipulation under anesthesia, and arthroscopic capsular release [2]. These treatments have all be shown to have short-term benefit in pain relief, but none have proven to be superior nor alter the long-term natural history of adhesive capsulitis.

Over the past decade, however, there has been a growing body of literature suggesting that Propionibacterium acnes infection may play a significant role in a variety of pathological conditions affecting the native shoulder, most notably frozen shoulder [4,5]. Our goal is to employ a treatment strategy focused on eradicating P acnes infection as a conservative treatment of adhesive capsulitis. Through this project, we aim to complete a prospective randomized pilot study to examine the hypothesis that administration of intra-articular antibiotics effective against P acnes will prove to be a superior treatment of adhesive capsulitis as compared to current gold standard of intraarticular steroid injection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older,
* diagnosis of stage II adhesive capsulitis as determined by clinical examination of the treating physician, and
* absence of abnormal findings on X-ray.

Exclusion Criteria:

* allergy to Doxycycline or Methylprednisolone,
* pregnancy,
* diagnosis,
* Inflammatory arthritis or diabetes,
* secondary adhesive capsulitis (history of significant trauma, rotator cuff tear injury, stroke)
* evidence of arthritis on x-ray,
* current infectious disease, and
* any previous treatment for the for adhesive capsulitis of the affected shoulder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E Kuhn, MD, Study Director — Study Director
Locations (1):
- Vanderbilt Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hsu JE, Anakwenze OA, Warrender WJ, Abboud JA. Current review of adhesive capsulitis. J Shoulder Elbow Surg. 2011 Apr;20(3):502-14. doi: 10.1016/j.jse.2010.08.023. Epub 2010 Dec 16. No abstract available. PMID 21167743
- [Result] Neviaser AS, Hannafin JA. Adhesive capsulitis: a review of current treatment. Am J Sports Med. 2010 Nov;38(11):2346-56. doi: 10.1177/0363546509348048. Epub 2010 Jan 28. PMID 20110457
- [Result] Hannafin JA, Chiaia TA. Adhesive capsulitis. A treatment approach. Clin Orthop Relat Res. 2000 Mar;(372):95-109. PMID 10738419
- [Result] Bunker TD, Boyd M, Gallacher S, Auckland CR, Kitson J, Smith CD. Association between Propionibacterium acnes and frozen shoulder: a pilot study. Shoulder Elbow. 2014 Oct;6(4):257-61. doi: 10.1177/1758573214533664. Epub 2014 May 27. PMID 27582943
- [Result] Levy O, Iyer S, Atoun E, Peter N, Hous N, Cash D, Musa F, Narvani AA. Propionibacterium acnes: an underestimated etiology in the pathogenesis of osteoarthritis? J Shoulder Elbow Surg. 2013 Apr;22(4):505-11. doi: 10.1016/j.jse.2012.07.007. Epub 2012 Sep 13. PMID 22981447
- [Result] Stirling A, Worthington T, Rafiq M, Lambert PA, Elliott TS. Association between sciatica and Propionibacterium acnes. Lancet. 2001 Jun 23;357(9273):2024-5. doi: 10.1016/S0140-6736(00)05109-6. No abstract available. PMID 11438138
- [Result] Dodson CC, Craig EV, Cordasco FA, Dines DM, Dines JS, Dicarlo E, Brause BD, Warren RF. Propionibacterium acnes infection after shoulder arthroplasty: a diagnostic challenge. J Shoulder Elbow Surg. 2010 Mar;19(2):303-7. doi: 10.1016/j.jse.2009.07.065. Epub 2009 Nov 1. PMID 19884021
- [Result] Athwal GS, Sperling JW, Rispoli DM, Cofield RH. Deep infection after rotator cuff repair. J Shoulder Elbow Surg. 2007 May-Jun;16(3):306-11. doi: 10.1016/j.jse.2006.05.013. Epub 2007 Feb 22. PMID 17321157
- [Result] Millett PJ, Yen YM, Price CS, Horan MP, van der Meijden OA, Elser F. Propionibacterium acnes infection as an occult cause of postoperative shoulder pain: a case series. Clin Orthop Relat Res. 2011 Oct;469(10):2824-30. doi: 10.1007/s11999-011-1767-4. Epub 2011 Jan 15. PMID 21240577
- [Result] Schneeberger AG, Yian E, Steens W. Injection-induced low-grade infection of the shoulder joint: preliminary results. Arch Orthop Trauma Surg. 2012 Oct;132(10):1387-92. doi: 10.1007/s00402-012-1562-z. Epub 2012 Jun 17. PMID 22707212
- [Result] Rollason J, McDowell A, Albert HB, Barnard E, Worthington T, Hilton AC, Vernallis A, Patrick S, Elliott T, Lambert P. Genotypic and antimicrobial characterisation of Propionibacterium acnes isolates from surgically excised lumbar disc herniations. Biomed Res Int. 2013;2013:530382. doi: 10.1155/2013/530382. Epub 2013 Aug 28. PMID 24066290
- [Result] Brandt KD, Mazzuca SA, Katz BP, Lane KA, Buckwalter KA, Yocum DE, Wolfe F, Schnitzer TJ, Moreland LW, Manzi S, Bradley JD, Sharma L, Oddis CV, Hugenberg ST, Heck LW. Effects of doxycycline on progression of osteoarthritis: results of a randomized, placebo-controlled, double-blind trial. Arthritis Rheum. 2005 Jul;52(7):2015-25. doi: 10.1002/art.21122. PMID 15986343
- [Result] Aydin O, Korkusuz F, Korkusuz P, Tezcaner A, Bilgic E, Yaprakci V, Keskin D. In vitro and in vivo evaluation of doxycycline-chondroitin sulfate/PCLmicrospheres for intraarticular treatment of osteoarthritis. J Biomed Mater Res B Appl Biomater. 2015 Aug;103(6):1238-48. doi: 10.1002/jbm.b.33303. Epub 2014 Oct 28. PMID 25350566
- [Result] Haerdi-Landerer MC, Suter MM, Steiner A. Intra-articular administration of doxycycline in calves. Am J Vet Res. 2007 Dec;68(12):1324-31. doi: 10.2460/ajvr.68.12.1324. PMID 18052736
- [Result] Cylwik J, Kita K, Barwijuk-Machala M, Reszec J, Klimiuk P, Sierakowski S, Sulkowski S. The influence of doxycycline on articular cartilage in experimental osteoarthrosis induced by iodoacetate. Folia Morphol (Warsz). 2004 May;63(2):237-9. PMID 15232785
- [Result] Bernal-Lagunas R, Aguilera-Soriano JL, Berges-Garcia A, Luna-Pizarro D, Perez-Hernandez E. Haemophilic arthropathy: the usefulness of intra-articular oxytetracycline (synoviorthesis) in the treatment of chronic synovitis in children. Haemophilia. 2011 Mar;17(2):296-9. doi: 10.1111/j.1365-2516.2010.02402.x. Epub 2010 Nov 11. PMID 21070486

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methylprednisolone | Doxycycline
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylprednisolone | Doxycycline | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in American Shoulder and Elbow Score (ASES)
Description: The American Shoulder and Elbow Score questionnaire was developed to provide a standardized method for evaluating shoulder function and has been validated in patients with any array of shoulder pathologies. ASES results are in the 0 to 100 range, where 0 indicates a worse shoulder condition and 100 indicates best shoulder condition, so the lower the score, the greater the level of shoulder disability. Transforming the pain and the ADLs domains into the final score relies on the following formulas: Pain = 5 x (10 - Score from question 7)
Time Frame: Baseline and 12 months
Population: 0 participants were analyzed due to the risk of de-identification with only 1 person enrolled.
Arm/Group | Methylprednisolone | Doxycycline
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Range of Motion(ROM) Measurements
Description: The ROM measurements will include forward flexion, abduction, external rotation at the side and at 90 degrees abduction, and internal rotation at the side and at 90 degrees abduction recorded by the treating physician at follow up visits
Time Frame: Baseline and 12 months
Population: 0 participants were analyzed due to the risk of de identification with only 1 person enrolled.
Arm/Group | Methylprednisolone | Doxycycline
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Medical Co-morbidities
Description: number of medical co-morbidities per participant
Time Frame: Baseline
Population: 0 parrticipants were ananlyzed due to the risk of de identification with only person enrolled.
Arm/Group | Methylprednisolone | Doxycycline
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Symptoms
Description: Length of time participants have experienced shoulder symptoms
Time Frame: Baseline
Population: 0 participants enrolled due to the risk of de identification with only 1 person enrolled.
Arm/Group | Methylprednisolone | Doxycycline
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Changes in Pain
Description: Number of participants with current dominant symptom and/or dominant symptom with disease onset
Time Frame: Baseline
Population: 0 participants enrolled due to the risk of de identifying with only 1 person enrolled.
Arm/Group | Methylprednisolone | Doxycycline
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pain With Sitting
Description: Number of patients that have pain while sitting or have ever had pain while sitting will be recorded using patient-reported survey and review of the patient's electronic medical record in Epic.
Time Frame: Baseline
Population: 0 participants enrolled due to the risk of de identifying with only 1 person enrolled.
Arm/Group | Methylprednisolone | Doxycycline
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Stiffness
Description: Number of participants with current dominant symptom and/or dominant symptom with disease onset
Time Frame: Baseline
Population: 0 participants enrolled due to the risk of de identifying with only 1 person enrolled
Arm/Group | Methylprednisolone | Doxycycline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: no patients were enrolled in the Doxycycline arm so the number at risk in that arm is zero.
Arm/Group | Methylprednisolone | Doxycycline
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT03479502/Prot_SAP_000.pdf